CLINICAL TRIAL: NCT06170606
Title: Prospective Multi-Site Safety and Effectiveness Study of the Boston Scientific Cardiac Cryoablation System for Drug Refractory, Recurrent Symptomatic Paroxysmal Atrial Fibrillation
Brief Title: POLARx Post Approval Study (POLARx PAS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PY008
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Cryoablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: prospective, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cryoablation (Experimental): Subjects undergoing cardiac ablation procedure with the Boston Scientific Cardiac Cryoablation System.
  Interventions: Device: Boston Scientific Cardiac Cryoablation System

INTERVENTIONS:
Device: Boston Scientific Cardiac Cryoablation System — The Boston Scientific Cardiac Cryoablation System is intended for ablation and electrical mapping of the pulmonary veins for pulmonary vein isolation (PVI) in the ablation treatment of patients with paroxysmal atrial fibrillation (PAF).The main devices and components of the system consists of the following:
  * POLARx™ or POLARx™ FIT Cryoablation Catheter
  * POLARMAP™ Catheter
  * POLARSHEATH™
  * SMARTFREEZE™ Console
  * Diaphragm Movement Sensor (DMS)
  * Related Accessories

SUMMARY:
To collect clinical data on safety, effectiveness and procedural success of Boston Scientific's Cardiac Cryoablation System (includes all BSC commercially available POLARx/POLARx Fit catheters) when used to perform pulmonary vein isolation (PVI) in the ablation treatment of de novo Atrial Fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

* Subjects indicated for drug refractory, recurrent symptomatic PAF treatment with the Cryoablation System, per physician's medical judgement, and as per standard of care
* Subjects who are willing and capable of providing informed consent;
* Subjects who are willing and capable of participating in all testing associated with this clinical study at an approved clinical investigational center;

Exclusion Criteria:

* Any known contraindication to an AF ablation or anticoagulation, including those listed in the IFU as legally approved conditions;
* Any prior LA ablation;
* Known or pre-existing severe PV Stenosis;
* Subjects with severe valvular disease OR with a prosthetic - mechanical or biological - heart valve (not including valve repair and annular rings);
* Presence of any pulmonary vein stents;
* Subjects with active systemic infection;
* Subject is unable or not willing to complete follow-up visits and examination for the duration of the study;- Subjects with life expectancy ≤ 1 year per investigator's medical judgement;
* Women of childbearing potential who are, or plan to become, pregnant during the time of the study (assessment per investigator's discretion);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Freedom From Primary Safety Events at 12 Months Post-procedure (Acute and Chronic Events) Using the Boston Scientific Cardiac Cryoablation System With POLARx Cryoablation Balloon Catheter Models | 12 Months
  This measure reports the observed safety event-free rate at 12 Months follow up for all treatment and intent subjects. The safety events are a composite of procedure-related and device-related adverse events. Acute Primary Safety Endpoints include:
  * Death
  * Myocardial infarction (MI)
  * Persistent gastroparesis/injury to vagus nerve
  * Transient ischemic attack (TIA)
  * Stroke/Cerebrovascular accident (CVA)
  * Thromboembolism/ Air embolism
  * Cardiac tamponade/perforation
  * Pneumothorax
  * Serious vascular access complications
  * Pulmonary edema/heart failure
  * AV block not attributable to medication effect or vasovagal reaction
  Chronic Primary Safety events (through 12 Months) include:
  * Atrial esophageal fistula
  * Pulmonary vein stenosis (≥ 70% reduction of diameter) OR presented by patient's symptoms at 12-Month follow-up and requiring intervention
Percentage of Participants With Freedom From Treatment Failure at 12 Months Post-procedure Using the Boston Scientific Cardiac Cryoablation System With POLARx Cryoablation Balloon Catheter Models | 12 Months
  This measure reports the observed failure-free rate at 12 Months post index procedure. Failure defined as:
  * Failure to achieve acute procedural success in the index procedure
  * Any documented recurrent AF episode(s), or new onset of AFL or AT events:
  * ≥ 30 seconds in duration from any clinical recording devices considered standard of care at the study center (excluding insertable loop recorders)or
  * ≥10-second of continuous AF, AFL or AT documented on any 12-lead ECG between Days 91 and 12-Month follow-up
  * Any of the following interventions for atrial fibrillation, or new onset of atrial flutter or atrial tachycardia between days 91 and 12 Month Follow Up:
  * Repeat procedure
  * Electrical and/or pharmacological cardioversion for AF/AFL/AT
  * Prescribed a higher dose of any AAD documented at baseline or a new AAD not documented at baseline.
  * Hospitalization for AF/AT/AFL

CONTACTS AND LOCATIONS:
Overall Officials: Wilber W Su, MD,FACC,FHRS, Study Chair — Banner- University Medical Group- Heart Center, Phoenix, AZ, USA
Locations (11):
- United States (11):
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Pima Heart & Vascular Clinical Research, Tucson, Arizona
  - Torrance Memorial Medical Center, Torrance, California
  - Intermountain Platte Valley Hospital, Brighton, Colorado
  - Valley View Hospital, Glenwood Springs, Colorado
  - St. Joseph's Hospital/BayCare Medical Group, Tampa, Florida
  - Bethesda North Hospital, Cincinnati, Ohio
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - University of Texas Medical Branch - Galveston, Galveston, Texas
  - Aurora Health, Grafton, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No requests for study data have been made at this time, however Boston's Scientific's policy on data sharing can be found at http://www.bostonscientific.com/en-US/data-sharing-requests.html